CLINICAL TRIAL: NCT00009256
Title: Analysis of HIV Genetic Variation in Patients Prior to Initiation of Highly Active Antiretroviral Therapy
Brief Title: Analysis of HIV Genetic Variation in Patients Before Beginning Highly Active Antiretroviral Therapy
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000110; 00-I-0110; NCT00005114 (obsolete NCT alias)
Record Dates: First submitted 2001-01-25; First posted 2001-01-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-03-03

CONDITIONS: HIV Infection
Keywords: Quasispecies Variation; Genotyping; Phenotyping; Antiretroviral Therapy; Drug Naive Patients; HIV; Treatment Naive
MeSH Terms: conditions — HIV Infections

SUMMARY:
The purpose of this study is to gain knowledge about why drug therapy sometimes stops working in people infected with the human immunodeficiency virus (HIV). This occurs in 30 to 40% of patients treated with powerful antiretroviral drugs. The study will examine how the virus becomes resistant to drug treatment through mutations (changes) and how different mutations produce new variants that are resistant to more than one drug.

HIV-infected patients 18 years and older who have not been treated with antiretroviral medications and who have a relatively stable amount of virus in their blood (viral load) may be eligible for this study. Pregnant or breastfeeding women may not participate. Candidates will be screened with blood tests to determine viral load and to study the genetics of the virus.

Participants will be hospitalized at the NIH Clinical Center for 10 days for daily blood sampling. (In exceptional circumstances, the sampling may be done on an outpatient basis.) After discharge, patients will be followed by weekly visits for blood tests for a total of 120 days. When antiretroviral treatment begins, the patient may do one of the following:

1. Continue on this study with antiretroviral treatment. Therapy will consist of D4T, 3TC, and efavirenz. Other drugs may be substituted for any of these that cannot be tolerated. HIV protease inhibitors will not be included in the regimen.
2. Complete participation in this study and, if eligible, enroll in another NIH protocol (AVBIO).
3. Begin standard antiretroviral therapy with a private physician.

Patients for whom treatment is not yet recommended or who choose not to be treated may continue to be monitored with blood tests for a total of 18 months. (Patients who leave the study after this time may re-join when they decide to start treatment.)

Participants may also undergo the following optional procedures to study the genetic variation of HIV: lymph node biopsy, spinal tap, and semen donation or female genital washing to collect secretion samples.

Sexual partners or needle-sharing partners of study patients are invited to enroll in this study to provide blood samples at the time the patient enrolls and at two intervals after any needle sharing or unsafe sex event they may report to NIH. Partners may also donate genital secretions or semen, and a lymph node or spinal fluid sample.

Information from this study may help in the development of new drug treatments that will be effective in controlling HIV infection when other treatments no longer work.

DETAILED DESCRIPTION:
Infection with human immunodeficiency virus (HIV) results in progressive immune destruction and death. Current therapy for HIV (highly active antiretroviral therapy or HAART) infection utilizes combinations of drugs that, under optimum conditions, inhibit HIV replication, halt progressive immunodeficiency, and permit a measure of immunological reconstitution. In its present form, however, HAART is inadequate. HAART does not cure HIV infection, and has significant adverse side effects, which may require drug discontinuation. One of the most challenging limitations of HAART is the development of drug resistance, which may occur in 30-40% of treated patients. The precise mechanisms responsible for drug resistance remain uncertain, but explanations include the emergence of HIV variants encoding genetic mutations that confer resistance to antiretroviral drugs. Such drug resistant mutations may occur and be present at low frequencies prior to drug therapy. Understanding how these mutations arise and remain circulating in populations of HIV is uncertain.

The purpose of the present protocol is to derive a comprehensive description of HIV population genetics in a longitudinal, observational study of HIV-infected patients prior to initiating antiretroviral therapy. We plan to utilize frequent blood sampling and an extensive sequencing strategy to investigate parameters of HIV population genetics, including: a) genotypic and phenotypic analyses of HIV drug resistance mutations, b) determinations of the rates at which mutations arise, become fixed, lost, or undergo recombination, c) linkage analyses, d) estimates of the size of the effective virus population. We plan to apply this information to develop models of HIV evolution, predict the genetic behavior of HIV populations, including the emergence of resistant genomes. We expect that information regarding HIV population genetics may assist in designing appropriate drug regimens to salvage control of HIV virus replication after initial regimens have failed.

ELIGIBILITY:
* INCLUSION CRITERIA:

HIV infection documented by ELISA/WB.

Viral load documented in our clinic as greater than or equal to 1000 copies RNA/ml plasma on one occasion.

At least 18 years of age.

For women of child-bearing potential, a negative serum pregnancy test is required within 14 days prior to enrollment.

Able to provide written informed consent.

EXCLUSION CRITERIA:

Absence of HIV infection within 8 weeks prior to entry, documented as a negative HIV ELISA and WB within 8 weeks of screening positive ELISA and WB.

Use of immunosuppressants or cytotoxic agents, with the exception of corticosteroids.

Presence of active AIDS defining opportunistic infection or malignancy requiring cytotoxic chemotherapy. Malignancies which do not require systemic cytotoxic chemotherapy, such as low grade non-progressive KS, or skin cancer treated with excision are not exclusion criteria.

Prior antiretroviral therapy with nucleoside or non-nucleoside RT inhibitors or protease inhibitors defined as: any therapy in the last 5 years; any more than 4 days of protease inhibitors or NNRTIs ever taken; any more than 2 weeks of NRTIs ever taken.

Psychiatric illness that in the opinion of the PI might interfere with study compliance.

Active substance abuse or history of prior substance abuse that may interfere with protocol compliance or compromise patient safety.

Refusal to practice safer sex practices or use precautions to prevent pregnancy (effective barrier birth control or abstinence).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65
Dates: Start 2000-04-13; Study Completion 2009-03-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Barrie KA, Perez EE, Lamers SL, Farmerie WG, Dunn BM, Sleasman JW, Goodenow MM. Natural variation in HIV-1 protease, Gag p7 and p6, and protease cleavage sites within gag/pol polyproteins: amino acid substitutions in the absence of protease inhibitors in mothers and children infected by human immunodeficiency virus type 1. Virology. 1996 May 15;219(2):407-16. doi: 10.1006/viro.1996.0266. PMID 8638406
- [Background] Birk M, Sonnerborg A. Variations in HIV-1 pol gene associated with reduced sensitivity to antiretroviral drugs in treatment-naive patients. AIDS. 1998 Dec 24;12(18):2369-75. doi: 10.1097/00002030-199818000-00005. PMID 9875574
- [Background] Butto S, Argentini C, Mazzella AM, Iannotti MP, Leone P, Leone P, Nicolosi A, Rezza G. Dual infection with different strains of the same HIV-1 subtype. AIDS. 1997 Apr;11(5):694-6. No abstract available. PMID 9108960